CLINICAL TRIAL: NCT03924206
Title: Hazardous Surgical Smoke: Risk Assessment and Evaluation of a New Smoke Extractor System (SES) in the Surgical Unit
Brief Title: Hazardous Surgical Smoke: Risk Assessment and Evaluation of a New Smoke Extractor System in the Surgical Unit
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Tofwerk AG, Thun Switzerland (equipment, data analysis) (Unknown); Lungenliga Bern (main funding) (Unknown); Erbe Swiss AG (equipment) (Unknown)
Responsible Party: Sponsor
Other Study IDs: SurgicalSmoke1
Record Dates: First submitted 2019-04-09; First posted 2019-04-23 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Lung Cancer; Lung Injury
Keywords: Smoke; Plume; Electrocautery; Mass spectrometer
MeSH Terms: conditions — Lung Neoplasms; Lung Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Minimally invasive surgery with smoke evacuation system (SES): minimally invasive surgical procedures during which a smoke evacuation device is used
  Interventions: Device: Smoke evacuation system
- Minimally invasive surgery without SES: minimally invasive surgical procedures during which no smoke evacuation device is used
- Open surgery with SES: open surgical procedures during which a smoke evacuation device is used
  Interventions: Device: Smoke evacuation system
- Open surgery without SES: open surgical procedures during which no smoke evacuation device is used

INTERVENTIONS:
Device: Smoke evacuation system — The smoke evacuation system removes the surgical smoke directly near the electrocautery tip, where it is generated
  Groups: Minimally invasive surgery with smoke evacuation system (SES); Open surgery with SES

SUMMARY:
The investigators will define two separate groups of surgical procedures: 1.) an 'open group' in which mainly open anatomic lung resections will be included, and 2.) a 'minimally invasive' group in which mainly thoracoscopic anatomic lung resections will be included.

Both groups will then be randomized to either the performance of the surgical procedure under 'standard conditions' or to the performance of the procedure with the additional use of a smoke evacuation system.

During every procedure the hazardous smoke that is generated by the electrocautery in the surgical field will be collected through a tube at the height of the surgeons face. The smoke is then directly transferred to a mass spectrometer that is situated in the operating room (OR) and performs a real-time analysis of the chemical substances in the air. The degree of air pollution will be measured as well as the smoke evacuation systems' ability to reduce these hazardous chemical substances in the air can be evaluated.

DETAILED DESCRIPTION:
Smoke samples will be continuously analyzed with a latest generation time of flight mass spectrometer in real time. Concerning the smoke evacuation device, the investigators will use the model IES 2 (Intelligent Evacuation System) from Erbe Swiss medical for this study.

Since this is only an observational study in which the investigators are only recording the type of surgery (i.e. open oder minimally invasive) and not recording sensitive patient data, the local ethics committee waived the need for an ethics committee approval of the study. In the end the smoke evacuation system does not have an effect on the patient or the procedure itself, but may rather influence the concentration of hazardous surgical fumes in the operating theatre.

ELIGIBILITY:
Inclusion Criteria:

- All surgical procedures with a planned duration of more than 1 hour

Exclusion Criteria:

* Patients with a contraindication for electrocautery use
* Patients with Pacemaker or implantable cardioverter-defibrillator (ICD)
* Patients with an implanted neurostimulator device

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All surgical procedures that will be performed during the study period at the investigators' department will be randomly allocated to either the performance of surgery with or the performance of surgery without the use of a mobile smoke evacuation device. Whether the procedure will be performed open or minimally invasive will be decided by the operating surgeon and is not part of the randomization process. During the respective surgeries, a mass spectrometer will be used to measure the smoke concentrations and its composition in the operating room.
Sampling Method: Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2019-09-09 (Actual)

PRIMARY OUTCOMES:
Hazardous fumes - specifically the concentration of Furfural, Benzene and Butadiene | assessment of measurement will start 4 months after the project is started and will take up to 12 weeks
  Analysis of surgical fume with real-time time of flight mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Gregor J Kocher, PD, MD, Principal Investigator — Division of Thoracic Surgery, University Hospital Bern, Switzerland
Locations (1):
- University Hospital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kocher GJ, Sesia SB, Lopez-Hilfiker F, Schmid RA. Surgical smoke: still an underestimated health hazard in the operating theatre. Eur J Cardiothorac Surg. 2019 Apr 1;55(4):626-631. doi: 10.1093/ejcts/ezy356. PMID 30388210
- [Derived] Kocher GJ, Koss AR, Groessl M, Schefold JC, Luedi MM, Quapp C, Dorn P, Lutz J, Cappellin L, Hutterli M, Lopez-Hilfiker FD, Al-Hurani M, Sesia SB. Electrocautery smoke exposure and efficacy of smoke evacuation systems in minimally invasive and open surgery: a prospective randomized study. Sci Rep. 2022 Mar 23;12(1):4941. doi: 10.1038/s41598-022-08970-y. PMID 35322134